CLINICAL TRIAL: NCT02383563
Title: Open-Label, Randomized, 24-Week Pilot Study of Metformin vs Observation for Persistent Immune Activation in Chronic HIV Infection
Brief Title: Metformin for HIV Inflammation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Hawaii (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H028; P30GM103341 (NIH)
Record Dates: First submitted 2015-02-09; First posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: HIV; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin Treatment Arm (Active Comparator): 500 mg metformin Extended Release tablets - one tablet daily increased at 4 weeks to 2 tablets (1000 mg) daily.
  Interventions: Drug: metformin extended release
- Observational Arm (No Intervention): Observation only

INTERVENTIONS:
Drug: metformin extended release
  Arms: Metformin Treatment Arm

SUMMARY:
This proposal seeks to assess the impact of 24 weeks of metformin on non-calcified plaques and calcified plaques assessed by coronary CT angiography, and on whether these changes can be explained by metformin-induced phenotypic and secretory changes of monocytes.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* on suppressive ART stable for > 1 year
* Age > 45 years
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Uncontrolled chronic medical condition or cancer
* Acute illness within 2 weeks of entry
* Diagnosis of diabetes or impaired fasting glucose
* Chronic diarrhea
* Known hypersensitivity or contraindication to metformin use
* Hepatitis C co-infection
* Serum B12 level below the reference normal range as listed by the commercial laboratory (Diagnostic Laboratory Services)
* Pregnancy, or intent to become pregnant
* Any immunomodulator, HIV vaccine, any other vaccine, or investigational therapy within 30 days of study entry.
* Current or past history of coronary artery disease or congestive heart failure
* Resting heart rate > 100 beats/min
* Presence of conduction abnormalities or pathologic arrhythmia on EKG
* The following lab values: Hemoglobin < 9.0 g/dL; Absolute neutrophil count < 1000/μL; Platelet count < 50,000/μL; and AST (SGOT) and ALT (SGPT) > 5x ULN
* Calculated creatinine clearance (Cockcroft and Gault) < 60 ml/min
* Patients over 450 lbs
* History of iodine allergy or X-ray contrast allergy
* History of allergy to metoprolol
* Active or recent past history (within past 2 years) of illicit substance or alcohol use or abuse which, in the judgment of the Investigator, will interfere with the patient's ability to comply with the protocol requirements
* Patients in whom there are other reasons that the CAC/CTA procedure is contra-indicated or who are at higher risk of adverse events
* Patients, who, in the opinion of the Investigator, are unable to comply with the dosing schedule and protocol evaluation or for whom the study may not be advisable

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Coronary plaques by CT angiography | 24 weeks
  change in total numbers of atherosclerotic plaques detected in the coronary arteries

SECONDARY OUTCOMES:
Monocyte subsets by multiparametric flow cytometry | 24 weeks
  change in numbers (cells/microliter of blood) of each monocyte subset (classical, intermediate, non-classical and transitional subsets)
Monocyte secretory function by intracellular cytokine staining release assay | 24 weeks
  Change in percent of monocytes secreting cytokine TNFalpha, percent secreting cytokine IL-6 and percent secreting cytokine IL-1beta
Sub-types of coronary plaques by CT angiography | 24 weeks
  Change in numbers of non-calcified atherosclerotic plaques detected in the coronary arteries; change in numbers of mixed plaques; change in numbers of calcified coronary plaques

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia M Shikuma, MD, Principal Investigator — University of Hawaii
Locations (1):
- Hawaii Center for AIDS, Honolulu, Hawaii, United States